CLINICAL TRIAL: NCT03930238
Title: VA MapTrek, an M-Health Intervention to Increase Steps Per Day in Rural Veterans
Brief Title: Increasing Steps Per Day in Rural Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Philip Polgreen, Professor of Medicine, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201901762
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Overweight
Keywords: Veterans
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA MapTrek (Experimental): Veterans in the intervention group receive a Fitbit and access to VA MapTrek, an interactive text-messaging platform. The only equipment needed is a Fitbit (we provide) and a smartphone (required to enroll). Each week, Veterans are assigned to a virtual walking route. Each day, they receive a text message with a link to the current route. The link will take them to a map where they can see their progress and the progress of others. A leaderboard provides information on how many steps each participant has taken. Throughout each race, participants will randomly receive challenge text messages. Completing a challenge awards bonus steps to propel their character along the map.
  Interventions: Behavioral: VA MapTrek
- Fitbit Only (Active Comparator): Veterans randomized to the control group will receive a Fitbit only. This will allow us to determine if changes in physical activity are due to VA MapTrek or simply by giving the Veterans a Fitbit.
  Interventions: Behavioral: Fitbit Only

INTERVENTIONS:
Behavioral: VA MapTrek — The objective is to report activity levels in our virtual environment to Veterans, thereby encouraging them to walk more.
  Arms: VA MapTrek
Behavioral: Fitbit Only — Fitbit Only
  Arms: Fitbit Only

SUMMARY:
VA MapTrek is a mobile-phone-based web application that allows participants to take a virtual walk in interesting locations around the world while tracking their progress against the progress of other veterans on an interactive map. Steps are counted using a commercially-available triaxial accelerometer (e.g., Fitbit), and users see their progress overlaid on Google Maps. The objective of this study is to report activity levels to veterans, thereby encouraging them to walk more. Once participants know how to text and use Google maps, no additional training is needed. VA MapTrek does not require a special app, so there are no logins or passwords to remember. Simply registering one's Fitbit and mobile phone at an initial enrollment meeting suffices.

DETAILED DESCRIPTION:
All consented participants will be provided with a Fitbit and instructed to wear it all day, every day for the next 9 weeks (The first few participants may require an additional week or two of wear as we will not begin the first MapTrek race until we have at least 5 participants enrolled in the study. They will be told this upon enrollment.). The enrollment process is expected to take anywhere from 15 to 45 minutes, depending on group assignment and participant familiarity with using Fitbits.

This, plus an exit survey (given via text message or phone, whichever the participant prefers), will be the extent of participation for the control group.

Members of the intervention group will be instructed on how to use MapTrek, the virtual walking race, and will also be given an instruction packet to refer to later. Data collected during the first week from the Fitbit will be used to compute baseline activity level. This baseline data will be used to place participants into an appropriate initial race group. Participants are placed into groups with other individuals who are active at a similar level, so that groups will be competitive.

Each virtual walking race will begin on Monday morning and end on Saturday night. Results of each race will be announced on Sundays. Depending on their performance each week, group assignment may change. Participants will compete in 8 week-long races over the course of the study.

Participants will receive 2-4 text messages per day including a daily status report and a link to view the race. They will also periodically receive challenge messages. If a participant completes a challenge, they will be awarded bonus steps to help move them along the route quicker.

To win a race, a participant must be furthest along on the route at 11:59 pm on Saturday. There is a leaderboard within MapTrek that helps participants determine their standing within each race. Participants are allowed to choose the screen name displayed on the leaderboard so that they may remain anonymous if desired.

At baseline, the following data will be collected about all participants: first and last name, last 4 of social security number (for consent documentation and to look up records in CPRS), age, sex, race, ethnicity, marital status, height, weight, body mass index, blood pressure, zip code, current medications, and comorbidities.

At the end of the study (9 weeks), the following data will be collected about all participants: height, weight, body mass index, blood pressure, current medications, and comorbidities.

At the end of the study (9 weeks), participants will be contacted via text message or phone call (based on their preference at baseline) to complete an exit survey. This survey will take approximately 10 minutes to complete. All participants will be contacted up to 3 times to complete the exit survey. If they cannot be reached, they will be considered lost to follow up.

ELIGIBILITY:
Inclusion Criteria:

* Comfortable speaking and reading in English
* BMI greater than or equal to 25
* Have a smart phone with texting and internet capabilities
* Willing to download the Fitbit app on their phone
* Must be a VA patient

Exclusion Criteria:

* Pregnancy
* Active mental health conditions that prevent them from providing consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Polgreen, MD, MPH, Principal Investigator — University of Iowa
Locations (1):
- VA Health Care System, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VA MapTrek | Fitbit Only
Started | 153 | 123
Collected Any Fitbit Data During Baseline Period | 152 | 114
Completed | 149 | 102
Not Completed | 4 | 21

BASELINE CHARACTERISTICS:
Population: All Veterans enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | VA MapTrek | Fitbit Only | Total
Number analyzed (Participants) | 153 | 123 | 276
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: 1 Veteran was older than 89 years of age, so their exact age could not be specified. 1 Veteran's age was missing.
  Years
    number analyzed (Participants) | 151 | 123 | 274
    (all) | 59.9 (12.7) | 61.9 (13.0) | 60.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 130 | 111 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 147 | 118 | 265
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 10 | 4 | 14
  White | 136 | 114 | 250
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 153 | 123 | 276
Lives in Urban Area [Count of Participants; unit: Participants] — Population: Address could not be determined for 1 Veteran in the Fitbit Only Group.
  Participants
    number analyzed (Participants) | 153 | 122 | 275
    (all) | 77 | 55 | 132
Marital Status [Count of Participants; unit: Participants]
  Currently Married | 113 | 83 | 196
  Previously Married | 31 | 29 | 60
  Never Married | 5 | 4 | 9
  Other | 4 | 7 | 11
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Missing participants did not have BMI values present in their medical record.
  kg/m^2
    number analyzed (Participants) | 152 | 121 | 273
    (all) | 32.9 (5.6) | 33.7 (5.8) | 33.2 (5.7)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Missing values were due to missing systolic blood pressures in the medical record.
  mmHg
    number analyzed (Participants) | 152 | 121 | 273
    (all) | 130.1 (14.6) | 130.0 (79.1) | 130.0 (14.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Missing values due to missing diastolic blood pressure values in the medical record.
  mmHg
    number analyzed (Participants) | 152 | 121 | 273
    (all) | 79.1 (8.2) | 79.1 (9.3) | 79.1 (8.7)
Number of Medications [Mean (Standard Deviation); unit: Medications] | 9.6 (6.9) | 9.4 (5.7) | 9.5 (6.4)
Number of Comorbidities [Mean (Standard Deviation); unit: Comorbidities] | 9.7 (5.9) | 10.3 (5.4) | 10.0 (5.7)
Days with Step Data [Mean (Standard Deviation); unit: Days] | 6.9 (5.0) | 4.6 (1.8) | 5.9 (4.2)
Number of Steps per Day [Mean (Standard Deviation); unit: Steps] — Population: Missing values due to Veterans not syncing Fitbit steps during baseline period.
  Steps
    number analyzed (Participants) | 147 | 108 | 255
    (all) | 7023 (4080) | 6754 (3545) | 6909 (3857)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Steps Per Day
Description: The Fitbit will provide the total number of steps that each Veteran has taken per day.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: Steps per day
Arm/Group | VA MapTrek | Fitbit Only
Number analyzed (Participants) | 149 | 102
Steps per day | 8756 (6251) | 7334 (4596)
Statistical Analysis 1: Comparison: VA MapTrek vs Fitbit Only; Test type: Superiority; Bayesian linear mixed effects regression — We did perform a Bayesian analysis which provided a posterior probability of 99.76% that the daily mean steps in the intervention group exceeded the daily mean steps in the comparison group; Group effect from Bayesian linear mixed = 1646 — Posterior standard deviation = 578. We have 95% credible intervals - the interval that contains 95% of the posterior probability distribution of the parameter of interest - which ranges from 511 to 2781

2. Secondary Outcome: Challenge Effectiveness
Description: Percentage of challenges that were met will be assessed.
Time Frame: 9 weeks
Population: Percentage of challenges met.
Measure: Number; unit: Percentage of Challenges Met
Units Other Than Participants: Challenges
Arm/Group | VA MapTrek
Number analyzed (Participants) | 153
Number analyzed (Challenges) | 3842
Percentage of Challenges Met | 2008
Statistical Analysis 1: Comparison: VA MapTrek; Test type: Other; Percentage = 53.3

3. Other Pre Specified Outcome: Completion of an Exit Survey
Description: Veterans will respond to an exit survey about their experiences with the study.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VA MapTrek | Fitbit Only
Number analyzed (Participants) | 153 | 123
Participants | 100 | 55

ADVERSE EVENTS:
Time Frame: 9 Weeks
Arm/Group | VA MapTrek | Fitbit Only
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/123
Other Adverse Events (participants affected / at risk) | 0/153 | 0/123

LIMITATIONS AND CAVEATS:
We do not know if Veterans wore the Fitbit or not. Days with partial wear will undercount total number of steps. However, this should be balanced between groups. Additionally, the groups were not equal because we had to stop enrollment early due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT03930238/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT03930238/SAP_001.pdf